CLINICAL TRIAL: NCT02749032
Title: Feed-Back Suppression of Meal-Induced GLP-1 Secretion Mediated Through Elevations in Intact GLP-1 Caused by Dipeptidyl Peptidase 4 (DPP-4) Inhibition: A Randomized, Prospective Comparison of Sitagliptin and Vildagliptin Treatment
Brief Title: Feed-Back Suppression of Meal-Induced Glucagon-like Peptide 1 (GLP-1) Secretion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michael A. Nauck (Other)
Responsible Party: Sponsor-Investigator, Michael A. Nauck, Prof. Dr. med. Michael A. Nauck, Diabeteszentrum Bad Lauterberg im Harz
Organization: Diabeteszentrum Bad Lauterberg im Harz (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DZBL-2010-1
Record Dates: First submitted 2016-04-08; First posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; Sitagliptin Phosphate; Metformin; Diet; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Vildagliptin - stratum diet/exercise (Active Comparator): Vildagliptin (50 mg per tablet) was administered orally twice daily (15 minutes prior to breakfast or test meal, on the last day of treatment period) and without a defined temporal relation to dinner in the evening, irrespective of the stratum defined by the background diabetes treatment.
  Mixed meal test were performed in the morning after an overnight fast.
  Interventions: Other: Mixed meal test; Drug: Vildagliptin; Other: Diet and exercise
- Vildagliptin - stratum metformin (Active Comparator): Vildagliptin (50 mg per tablet) was administered orally twice daily (15 minutes prior to breakfast or test meal, on the last day of treatment period) and without a defined temporal relation to dinner in the evening, irrespective of the stratum defined by the background diabetes treatment.
  Mixed meal test were performed in the morning after an overnight fast.
  Interventions: Other: Mixed meal test; Drug: Vildagliptin; Drug: Metformin
- Sitagliptin - stratum diet/exercise (Active Comparator): The dosage of sitagliptin depended on the stratum defined by the background diabetes medication. In patients treated with diet and exercise (no other glucose-.lowering medication), sitagliptin was given as one 100 mg in the morning (15 minutes prior to breakfast or the test meal, on the last day of the treatment period), and a corresponding placebo tablet was administered in the evening (no temporal relation to dinner required).
  Mixed meal test were performed in the morning after an overnight fast.
  Interventions: Other: Mixed meal test; Drug: Sitagliptin; Other: Diet and exercise
- Sitagliptin - stratum metformin (Active Comparator): In patients treated with metformin, sitagliptin (50 mg per tablet) was administered orally twice daily (15 minutes prior to breakfast or test meal, on the last day of treatment period) and without a defined temporal relation to dinner in the evening.
  Mixed meal test were performed in the morning after an overnight fast.
  Interventions: Other: Mixed meal test; Drug: Sitagliptin; Drug: Metformin
- Placebo - stratum diet/exercise (Placebo Comparator): Placebo was administered orally twice daily: 15 minutes prior to breakfast or the test meal on the last day of treatment period) and one dose in the evening (no temporal relation to dinner required).
  Mixed meal test were performed in the morning after an overnight fast.
  Interventions: Other: Mixed meal test; Drug: Placebo; Other: Diet and exercise
- Placebo - stratum metformin (Placebo Comparator): Placebo was administered orally twice daily: 15 minutes prior to breakfast or the test meal on the last day of treatment period) and one dose in the evening (no temporal relation to dinner required).
  Mixed meal test were performed in the morning after an overnight fast.
  Interventions: Other: Mixed meal test; Drug: Placebo; Drug: Metformin

INTERVENTIONS:
Other: Mixed meal test — Mixed meal test were performed in the morning after an overnight fast. The standardized mixed meal was composed of 2 eggs (100 g), 1 slice (50 g) of whole grain rye bread, 1 slice (50 g) of rye flour bread, 10 g of fat-reduced margarine, 20 g of boiled ham, and 25 g of diet jam, amounting to 450 kcal, 50 % carbohydrate, 20 % protein, and 30 % fat (based on calorie count). Patients were allowed to drink tea (black or fruit-based) or de-caffeinated coffee ad libitum.
Drug: Vildagliptin — Vildagliptin (50 mg per tablet) was administered orally twice daily (15 minutes prior to breakfast or test meal, on the last day of treatment period) and without a defined temporal relation to dinner in the evening, irrespective of the stratum defined by the background diabetes treatment.
  Arms: Vildagliptin - stratum diet/exercise; Vildagliptin - stratum metformin
Drug: Sitagliptin — The dosage of sitagliptin depended on the stratum defined by the background diabetes medication. In patients treated with diet and exercise (no other glucose-.lowering medication), sitagliptin was given as one 100 mg in the morning (15 minutes prior to breakfast or the test meal, on the last day of the treatment period), and a corresponding placebo tablet was administered in the evening (no temporal relation to dinner required).
  Arms: Sitagliptin - stratum diet/exercise; Sitagliptin - stratum metformin
Drug: Placebo — Placebo was administered orally twice daily: 15 minutes prior to breakfast or the test meal on the last day of treatment period) and one dose in the evening (no temporal relation to dinner required).
  Arms: Placebo - stratum diet/exercise; Placebo - stratum metformin
Drug: Metformin — For patients continuing with pre-existing metformin treatment, 1000 mg film coated tablets from commercial sources. In half of the patients (stratum: metformin as background medication), metformin was administered orally twice daily at 1000 mg of active compound during of after breakfast and dinner.
  Arms: Placebo - stratum metformin; Sitagliptin - stratum metformin; Vildagliptin - stratum metformin
Other: Diet and exercise — Patients treated their diabetes mellitus type 2 with diet/exercise only
  Arms: Placebo - stratum diet/exercise; Sitagliptin - stratum diet/exercise; Vildagliptin - stratum diet/exercise

SUMMARY:
The present study is a phase I, single-centre, double-blind, randomized, cross-over (3 treatments, 3 treatment periods and 6 sequences), stratified (background medication: metformin vs. diet-only), placebo-controlled study, comparing periods lasting 6-9 days on treatment with repeated doses of vildagliptin, sitagliptin, or placebo, with wash-out periods between treatment periods lasting 21 days minimum.

The study was designed to directly compare the effects of vildagliptin and sitagliptin on incretin hormone responses, glycaemia, and insulin as well as glucagon secretory responses in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Design. The present study is a phase I, single-centre, double-blind, randomized, cross-over (3 treatments, 3 treatment periods and 6 sequences), stratified (background medication: metformin vs. diet-only), placebo-controlled study, comparing periods lasting 6-9 days on treatment with repeated doses of vildagliptin, sitagliptin, or placebo, with wash-out periods between treatment periods lasting 21 days minimum.

Experimental procedures. Meal tests were performed in the morning after an overnight fast. The standardized mixed meal was composed of 2 eggs (100 g), 1 slice (50 g) of whole grain rye bread, 1 slice (50 g) of rye flour bread, 10 g of fat-reduced margarine, 20 g of boiled ham, and 25 g of diet jam, amounting to 450 kcal, 50 % carbohydrate, 20 % protein, and 30 % fat (based on calorie count). Patients were allowed to drink tea (black or fruit-based) or de-caffeinated coffee ad libitum.

Blood sampling. Plasma glucose was determined in capillary samples taken from hyperaemic ear lobes. Venous blood was collected from indwelling venous cannulas placed in a distal forearm vein, for the determination of insulin, C-peptide, glucagon, GLP-1 (total), GLP-1 (intact), glucose-dependent insulinotropic polypeptide (GIP) (total), GIP (intact), and free fatty acids. After drawing basal blood specimens at -15 and 0 min, blood was taken at 15, 30, 45, 60, 90, 120, 180, and 240 min.

Laboratory determinations. Glucose, insulin, C-peptide, total GLP-1 (C-terminally directed assay), intact GLP-1 (sandwich ELISA), total GIP (C-terminally directed assay), intact GIP (N-terminally directed assay) and glucagon were determined.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus type 2 for more than one year, as defined by the American Diabetes Association
* body-mass-index between 20.0 and 40.0 kg/m² (inclusive),
* glycohaemoglobin (HbA1c) ≤ 8.5%,
* normal vital signs after 10 minutes resting in the supine position: systolic blood pressure 96 mmHg -159 mmHg; diastolic blood pressure 46 mmHg-99 mmHg; heart rate 46-99 bpm
* laboratory parameters within the normal range, or abnormalities judged to be clinically irrelevant by the investigator (serum estimated glomerular filtration rate was enforced to be > 60 ml/min; hepatic enzymes and bilirubin (unless the subject has documented Gilbert syndrome) had to be > 3-fold the upper limit of normal)
* women of childbearing potential (less than two years post-menopausal or not surgically sterile for more than 3 months), had to prove a negative serum β-human chorionic gonadotropin (HCG) pregnancy test at screening and a negative urine β-HCG pregnancy test at day 1 on each of the treatment periods, had to use a highly effective method of birth control (failure rate less than 1% per year)
* normal or clinically irrelevant findings in medical history and physical examination

Exclusion Criteria:

* any glucose-lowering drug therapy other than metformin during 3 months before the first treatment period
* any history or presence of clinically relevant cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic (apart from diabetes mellitus type 2), haematological, neurological, psychiatric, systemic, ocular, gynaecologic, or infectious disease; any acute infectious disease or signs of acute illness
* symptoms of a clinically significant illness in the 3 months before the study, which, according to the investigator's opinion, could interfere with the purposes of the study
* congestive heart failure of New York Heart Association (NYHA) functional class III-IV
* Regular use of any medication other than metformin in the last month before study start with the exception of thyroid hormones, lipid-lowering and antihypertensive drugs, and, if female, with the exception of hormonal contraception or menopausal hormone replacement therapy
* blood loss (>300 ml, any reason) within 3 months before inclusion, or a haemoglobin < 11.0 g/dl
* participation in a trial with any investigational drug during the past three months
* presence or history of a drug allergy or clinically significant allergic disease according to the investigator's judgment including any known hypersensitivity to DPP-4 inhibitors
* presence of drug or alcohol abuse (alcohol consumption > 40 grams / day)
* if female, pregnancy (defined as positive β-HCG blood test), breast-feeding

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-11; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
GLP-1 feedback inhibition | 0-240 min following meal ingestion
  Comparison of the percentage reduction or its reciprocal value (times 100) in total GLP-1 (secretion, incremental values above baseline, 0-240 min following meal ingestion) between vildagliptin and sitagliptin treatment relative to placebo treatment.

SECONDARY OUTCOMES:
Relationship of the GLP-1 feedback inhibition [%] | 0-240 min following meal ingestion
  Relationship of the GLP-1 feedback inhibition [%] by DPP-4 inhibition to meal-related plasma responses of "total" and "intact" incretin hormone concentrations
Differences in glucagon secretion [pmol/l] | 0-240 min following meal ingestion
  Differences in glucagon secretion [pmol/l] between vildagliptin and sitagliptin treatment relative to placebo treatment during mixed meal tests
Differences in insulin secretory responses - Insulin [pmol/l] | 0-240 min following meal ingestion
  Differences in insulin secretory responses due to insulin concentration between vildagliptin and sitagliptin treatment relative to placebo [pmol/l] treatment during mixed meal tests
Differences in insulin secretory responses - c-peptide [pmol/l] | 0-240 min following meal ingestion
  Differences in insulin secretory responses due to c-peptide [pmol/l] concentration between vildagliptin and sitagliptin treatment relative to placebo treatment during mixed meal tests
Differences in glucose concentrations [mmol/l] | 0-240 min following meal ingestion
  Differences in glucose concentrations [mmol/l] between vildagliptin and sitagliptin treatment relative to placebo treatment during mixed meal tests
Incidence of Treatment-Emergent Adverse Events - Safety and tolerability | From date of screening until the end of study date, assessed for up to 4.7 months
  Safety and tolerability of treatments were assessed for A) period between screening visit and first treatment period (3 to 28 days),B) Three treatment periods 7 to 9 days each (21 - 28 days),C) 2 wash-out periods between 21 - 40 days (42 - 80 days), and D) Period between last treatment visit and end of study visit (1 day). In total that are 67 - 136 days (2.2 - 4.7 month). Patients were ask for any adverse events. Incidence of Treatment-Emergent Adverse Events were analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Nauck, Prof., Principal Investigator — Diabeteszentrum Bad Lauterberg
Locations (1):
- Diabeteszentrum Bad Lauterberg, Bad Lauterberg im Harz, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided